CLINICAL TRIAL: NCT05658783
Title: The Effect of Footbath on Pain Severity and Sleep Quality Levels of Patients With Lumbar Degenerative Disc Disease
Brief Title: Effect of Footbath on Pain Severity and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Seher Ünver, Associate Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-PO119
Record Dates: First submitted 2022-11-17; First posted 2022-12-21 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Foot; Sleep; Pain
Keywords: Footbath; Perioperative nursing; Post-operative pain; Sleep quality
MeSH Terms: conditions — Pain; Pain, Postoperative; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analysed by a independent researcher
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this study group will be asked to keep their feet in 42oC (42 Degrees Celsius) hot water for 20 minutes on the night of the day of surgery.
  Interventions: Other: Hot water foot bath
- Control Group (No Intervention): Participants in this study group will take the standard service clinical procedure and hot water foot bath will not be applied.

INTERVENTIONS:
Other: Hot water foot bath — Keeping keep in 42oC (42 Degrees Celsius) hot water for 20 minutes
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to examine the effect of hot water foot bath on the patients' pain severity and sleep quality levels on the night of the lumbar degenerative disc surgery. The main hypotheses are:

* H1=Pain severity of the patients who applied footbath is lower than the patients who did not.
* H2=The sleep quality of the patients who applied footbath is higher than the patients who did not.

Participants will be asked to keep their feet in 42oC hot water for 20 minutes on the night of the day of surgery.

If there is a comparison group: Researchers will compare control group to see if there is any difference on the pain severity and sleep quality of the patients.

DETAILED DESCRIPTION:
Group allocation of the patients was done through using Random Allocation Software program and patients were allocated into two groups: the intervention group and the control group.

Patients in the intervention group were asked to take a footbath in 42oC water for 20-minutes in the evening of the surgery day.

The nurse researcher visited the patients in the morning of the surgery day in their service room, asked to rate their current pain severity score between 0 - 10 points, and asked to rate the sleep quality scale items between 0 - 100 points according to their previous night sleep. The patients in the intervention group were informed that they were going to be visited to perform the footbath in the evening before they go asleep, and the patients in the control group were informed that they were going to be visited in the next morning.

In the evening of the surgery day, the nurse researcher visited the patients in their service room and explained footbath procedure to the patients, following, filled the foot tub with hot water to approximately 20 cm above the patients' ankle and measured the temperature of the water with using a water thermometer. When the temperature was stable at 42oC, the patients were asked to sit in semi-fowler position in the bed and to immerse their feet in the foot tub without washing or any massage for 20-minutes. During the footbath, the upper side of the foot tub was covered with a towel to prevent temperature loss by vaporizing and the researcher stayed in the room to observe the patient according to any unwanted events such as sweating, having pain, feeling hot or bad etc. At the end of the footbath procedure, feet of the patients were dried with a towel and checked for any redness. Then, the researcher helped patients to wear their socks to keep the feet warm and measured the final temperature of the water. Finally, the patients were informed that they were going to be visited in the morning.

The standard procedure is pharmacological pain management following the surgery as explained under the study setting title to decrease the pain severity, consequently, to improve the sleep quality, and this standard procedure was used for each group. Footbath was not applied to the patients in the control group.

Patients in both study groups were visited by the nurse researcher in the morning of the postoperative day in their service room, asked to rate their current pain severity score between 0 - 10 points, and asked to rate the sleep quality scale items between 0 - 100 points according to their previous night sleep.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Undergoing elective surgery
* Surgery planned for lumbar degenerative disc disease
* No known sleep problems and no sleeping pills
* Patients admitted to the ward at least 1 day before the operation
* Those who will spend the night of the day after the operation in the service
* Verbal communicative
* Those who want to take a foot bath in 42oC water

Exclusion Criteria:

* Younger than 18 years old
* Unplanned surgery
* Have a diagnosed sleep problem and using sleeping pills
* Having communication problems
* Not volunteering to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Pain severity | In the morning of the surgery day and in the morning of the post-operative day
  will be evaluated with using the Visual Analog Scale (VAS), between "0-no pain" score and "10-unbearable pain" score, is used to evaluate perceived back and/or leg pain severity.
Sleep quality | In the morning of the surgery day and in the morning of the post-operative day
  will be evaluated with using the Visual Analog Sleep Scale (VAS-Scale), numbers ranging from 0 (left side) to 100 (right side), is used to evaluate the previous night's sleep quality of patients. This scale was developed by Verran and Snyder-Halpern and the Turkish validity and reliability of the scale was completed by Çetinkaya and Karabulut. It has one dimension and 10 items.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Ünver, Principal Investigator — Trakya University; Ülkü Çolakoğlu, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Seher Ünver, Edirne
  - Başakşehir Çam and Sakura City Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided